CLINICAL TRIAL: NCT00816400
Title: A Phase 1, Multicenter, Open-label, Single-arm, Dose-escalation Study to Evaluate the Safety, Tolerability, and Antitumor Activity of MEDI-575, a Fully Human Monoclonal Antibody Directed Against Platelet-derived Growth Factor Receptor Alpha (PDGFRα), in Subjects With Advanced Solid Tumors Refractory to Standard Therapy or for Which No Standard Therapy Exists
Brief Title: A Dose Escalation, Dose Expansion Study to Evaluate the Safety, Tolerability, and Antitumor Activity of MEDI-575, in Subjects With Advanced Tumors.
Acronym: MEDI-575
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP187
Record Dates: First submitted 2008-12-23; First posted 2009-01-01 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Tovetumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) (Experimental): Single lead-in dose of MEDI-575 at 0.5 mg/kg as a 60-minute intravenous (IV) infusion administered 7 days prior to first dose at 3.0 mg/kg; MEDI-575 administered at 3.0 mg/kg as a 60-minute IV infusion on Study Days 1, 8, and 15 (once every 7 days [QWk]) of each 21-day treatment cycle until unacceptable toxicity, documentation of disease progression, or other reasons for participant withdrawal occurred.
  Interventions: Drug: MEDI-575
- MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) (Experimental): MEDI-575 administered at 6.0 mg/kg as a 60-minute IV infusion on Study Days 1, 8, and 15 (QWk) of each 21-day treatment cycle until unacceptable toxicity, documentation of disease progression, or other reasons for participant withdrawal occurred.
  Interventions: Drug: MEDI-575
- MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) (Experimental): MEDI-575 administered at 9.0 mg/kg as a 60-minute IV infusion on Study Days 1, 8, and 15 (QWk) of each 21-day treatment cycle until unacceptable toxicity, documentation of disease progression, or other reasons for participant withdrawal occurred.
  Interventions: Drug: MEDI-575
- MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) (Experimental): MEDI-575 administered at 12.0 mg/kg as a 60-minute IV infusion on Study Days 1, 8, and 15 (QWk) of each 21-day treatment cycle until unacceptable toxicity, documentation of disease progression, or other reasons for participant withdrawal occurred.
  Interventions: Drug: MEDI-575
- MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) (Experimental): MEDI-575 administered at 15.0 mg/kg as a 60-minute IV infusion on Study Days 1, 8, and 15 (QWk) of each 21-day treatment cycle until unacceptable toxicity, documentation of disease progression, or other reasons for participant withdrawal occurred.
  Interventions: Drug: MEDI-575
- MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) (Experimental): MEDI-575 administered at 25.0 mg/kg as a 90-minute IV infusion on Study Day 1 of each 21-day treatment cycle (once every 21 days [Q3Wk]) until unacceptable toxicity, documentation of disease progression, or other reasons for participant withdrawal occurred.
  Interventions: Drug: MEDI-575
- MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) (Experimental): MEDI-575 administered at 35.0 mg/kg as a 90-minute IV infusion on Study Day 1 of each 21-day treatment cycle (Q3Wk) until unacceptable toxicity, documentation of disease progression, or other reasons for participant withdrawal occurred.
  Interventions: Drug: MEDI-575
- MEDI-575, 9.0 mg/kg QWk Expansion Phase (Experimental): MEDI-575 administered at 9.0 mg/kg as a 60-minute IV infusion on Study Days 1, 8, and 15 (QWk) of each 21-day treatment cycle until unacceptable toxicity, documentation of disease progression, or other reasons for participant withdrawal occurred.
  Interventions: Drug: MEDI-575
- MEDI-575, 25 mg/kg Q3Wk Expansion Phase (Experimental): MEDI-575 administered at 25.0 mg/kg as a 90-minute IV infusion on Study Day 1 of each 21-day treatment cycle (Q3Wk) until unacceptable toxicity, documentation of disease progression, or other reasons for participant withdrawal occurred.
  Interventions: Drug: MEDI-575

INTERVENTIONS:
Drug: MEDI-575 — MEDI-575 as an IV infusion

SUMMARY:
Evaluate the safety, tolerability and the tolerated maximum dose of MEDI-575 in adult subjects with advanced solid tumors refractory to standard therapy or for which no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumor for which no curative or standard therapies exist
* Karnofsky performance status of ≥ 60
* Life expectancy of >12 weeks
* Adequate hematologic and organ function
* Negative serum pregnancy test (women only)
* Two methods of birth control for female participants of child-bearing potential or male participants with their female partners of child-bearing potential

Exclusion Criteria:

* Prior chemotherapy or investigational treatment within 4 weeks of study drug administration
* Prior biological or immunological treatment within 6 weeks of study drug administration
* Concurrent therapy for of cancer
* Major surgery within four weeks or minor surgery within two weeks of study drug administration
* History of diabetes or current treatment for diabetes
* New York Heart Association ≥ Grade 2 congestive heart failure
* History of myocardial infarction, unstable angina, transient ischemic attack or stroke within the previous 6 months prior to study entry
* History of other invasive malignancy within 5 years (exceptions are cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that are surgically cured)
* Significant active infection
* Known brain metastases
* Pregnancy or lactation or plans to become pregnant while on study
* Clinically significant abnormality on ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-03-02 (Actual); Primary Completion 2012-01-19 (Actual); Study Completion 2012-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Denver, Colorado
  - Research Site, Indianapolis, Indiana
  - Research Site, Las Vegas, Nevada
  - Research Site, Dallas, Texas
  - Research Site, Norfolk, Virginia

REFERENCES:
- [Background] Becerra CR, Conkling P, Vogelzang N, Wu H, Hong S, Narwal R, Liang M, Tavakkoli F, Pandya N. A phase I dose-escalation study of MEDI-575, a PDGFRalpha monoclonal antibody, in adults with advanced solid tumors. Cancer Chemother Pharmacol. 2014 Nov;74(5):917-25. doi: 10.1007/s00280-014-2567-9. Epub 2014 Aug 23. PMID 25149088
- See also: MEDI-575_CP-187_Protocol_Redacted_28Aug14 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=19&filename=MEDI-575_CP-187_Protocol_Redacted_28Aug14.pdf
- See also: PMCID: PMC3749129: Circulating Tumor Cells: Application as a Biomarker for Molecular Characterization and Predictor of Survival in an All-Comer Solid Tumor Phase I Clinical Study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3749129/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 5 centers in the United States between March 2009 and January 2012.
Pre-assignment Details: A total of 49 participants were screened, out of these, 35 participants were randomized.
Period: Overall Study
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Started | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 6 | 6
Completed | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not Completed | 2 | 3 | 5 | 3 | 2 | 3 | 2 | 5 | 6
Not completed — Death | 2 | 3 | 3 | 3 | 2 | 3 | 2 | 5 | 6
Not completed — In hospice care at the end of the study | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase | Total
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 6 | 6 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (16.5) | 65.0 (8.5) | 60.2 (8.5) | 66.3 (9.1) | 67.0 (10.5) | 58.0 (8.5) | 68.3 (8.4) | 68.2 (15.1) | 59.3 (6.6) | 63.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 2 | 2 | 1 | 0 | 3 | 3 | 16
  Male | 2 | 0 | 4 | 1 | 1 | 2 | 3 | 3 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. Treatment-emergent AEs (TEAEs) are events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug, for the period extending to 30 days after the last dose of study drug. Participants were counted only once for each event and by the highest event severity, regardless of how many events the participant experienced. The AEs were summarized using Medical Dictionary for Regulatory Activities (MedDRA) version 14.1.
Time Frame: From the start of study drug administration through 30 days after last dose of MEDI-575, up to 112 weeks
Population: Safety population: All participants who have received any treatment of MEDI-575
Measure: Number; unit: Participants
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 6 | 6
Participants | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 6 | 6

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: A serious AE (SAE) is any AE that results in death, is immediately life threatening, require (or prolong) inpatient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, or is an important medical event that may jeopardize the participant or may require medical intervention to prevent one of the outcomes listed above. Treatment-emergent SAEs that emerged after start of study drug were reported. Participants were counted only once for each event and by the highest event severity, regardless of how many events the participant experienced. The SAEs were summarized using MedDRA version 14.1.
Time Frame: From the start of study drug administration through 30 days after last dose of MEDI-575, up to 112 weeks
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 6 | 6
Participants | 0 | 1 | 3 | 0 | 0 | 1 | 2 | 5 | 1

3. Primary Outcome: Treatment-emergent Adverse Events Related to Laboratory Parameters
Description: Laboratory evaluations of blood and urine samples were performed, including hematology (complete blood count, differential, and platelet count); serum chemistry (SrChem) aspartate transaminase (AST), alanine transaminase, total bilirubin, creatinine, alkaline phosphatase, sodium, potassium, chloride, phosphorus, calcium, glucose, magnesium, albumin, and lactate dehydrogenase); and routine urinalysis. Number of participants with TEAEs related to laboratory evaluations were reported.
Time Frame: From the start of study drug administration through 30 days after last dose of MEDI-575, up to 112 weeks
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 6 | 6
Participants
  Hematology: Anaemia | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2
  Hematology: Leukocytosis | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Hematology: Thrombocytopenia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  SrChem: AST increased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  SrChem: Blood Alkaline phosphatase increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  SrChem: Blood creatinine increased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  SrChem: Hypercalcaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  SrChem: Hyperglycaemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  SrChem: Hyperkalaemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  SrChem: Hypokalaemia | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 1 | 1
  SrChem: Hypomagnesaemia | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
  SrChem: Hyponatraemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  SrChem: Hypophosphataemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Urinalysis: Urine colour abnormal | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urinalysis:Urobilinogen urine increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Urinalysis:Haematuria | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urinalysis:Proteinuria | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Treatment-emergent Adverse Events Related to Electrocardiogram Evaluations
Description: All 12-lead electrocardiograms (ECGs) performed during the study were obtained in triplicate (ie, 3 ECGs were obtained within a 5-minute time interval) and analyzed. ECG parameters included heart rate (high and low), QT interval, QTcB (corrected QT interval per Bazett's formula), and QTcF (corrected QT interval per Fridericia's formula). Number of participants with TEAEs related to ECG after the start of study drug were reported.
Time Frame: From the start of study drug administration through 30 days after last dose of MEDI-575, up to 112 weeks
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 6 | 6
Participants
  Supraventricular tachycardia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Tachycardia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0

5. Primary Outcome: Treatment-emergent Adverse Events Related to Vital Sign Parameters
Description: Vital signs (temperature, blood pressure, pulse rate, and respiratory rate) were performed throughout the study. The TEAEs related to vital signs in participants were reported.
Time Frame: From the start of study drug administration through 30 days after last dose of MEDI-575, up to 112 weeks
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 6 | 6
Participants
  Pyrexia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypertension | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Hypotension | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

6. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: For the dose escalation phase, a minimum of 21 evaluable participants (3 participants each in Dose Cohorts 1 through 7) were required for this study if Dose Limiting Toxicities (DLTs) do not occur. If a DLT does occur among the first 3 participants in a cohort, 3 additional participants were to be added to the cohort; 3 more participants were to be added to a cohort to determine the MTD if only 3 participants have been previously treated at that dose. The MTD is the maximum dose at which no more than 1 out of 6 participants experienced a DLT. A DLT is defined as any grade 3 or higher hematologic toxicity or any grade 3 or higher non-hematologic toxicity except grade 3 fever (in the absence of neutropenia) or grade 3 rigors/chills.
Time Frame: From the start of study drug administration through 30 days after last dose of MEDI-575, up to 112 weeks
Population: MTD evaluable population includes all participants in the dose escalation phase who have received at least 1 full cycle of MEDI-575 and have completed the safety follow-up through the DLT-evaluation period, or who experienced a DLT. The MTD dose was not evaluated as there were no DLTs reported in this study.
Measure: Number; unit: Milligrams per kilogram (mg/kg)
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7)
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 3 | 3
Milligrams per kilogram (mg/kg) | NA — There are no observations for this Table | NA — There are no observations for this Table | NA — There are no observations for this Table | NA — There are no observations for this Table | NA — There are no observations for this Table | NA — There are no observations for this Table | NA — There are no observations for this Table

7. Secondary Outcome: Pharmacokinetics (PK) of MEDI-575 After the First Dose: Observed Maximum Serum Concentration (Cmax)
Description: The concentration of MEDI-575 quantitatively determined in serum samples using a validated electrochemiluminescence (ECL) PK assay. The Cmax after the first dose was obtained directly from the measured concentration-time curves. The concentration-time curve is the result of blood sampling at specified time points and its measured concentration of MEDI-575.
Time Frame: For 0.5/3, 6, 9, 12, 15 mg/kg: Cycle 1: Day 1 (pre- and end of infusion, 2 and 6 hours post infusion), Days 2, 3 and 8 (pre-dose); For 25 and 35 mg/kg: Cycle 1: Day 1 (pre- and end of infusion, 2 and 6 hours post infusion), Days 2, 3, 8 and 15.
Population: All the participants who received first dose of MEDI-575 and for whom PK blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter (μg/mL)
Groups:
- MEDI-575, 0.5 mg/kg QWk Escalation Phase (Cohort 1): Single lead-in dose of MEDI-575 at 0.5 mg/kg as a 60-minute intravenous (IV) infusion administered 7 days prior to first dose at 3.0 mg/kg
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 0.5 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 3 | 6 | 6
Micrograms per milliliter (μg/mL) | 72.6 (7.00) | 154 (44.9) | 239 (98.1) | 590 (124) | 632 (20.0) | 670 (131) | 918 (111) | 10.9 (0.512) | 240 (44.1) | 549 (143)

8. Secondary Outcome: PK of MEDI-575 After the First Dose: Time to Maximum Concentration (Tmax)
Description: The time to reach maximum serum concentration after the first dose of MEDI-575 was obtained directly from the measured concentration-time curves. The concentration-time curve is the result of blood sampling at specified time points and its measured concentration of MEDI-575.
Time Frame: as for outcome 7
Population: All the participants who received first dose of MEDI-575 and for whom PK blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 0.5 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 3 | 6 | 6
Day | 0.0759 (0.0545) | 0.0479 (0.00318) | 0.0618 (0.0381) | 0.130 (0.142) | 0.106 (0.0381) | 0.227 (0.142) | 0.0639 (0.00139) | 0.103 (0.0498) | 0.139 (0.0804) | 0.118 (0.0941)

9. Secondary Outcome: PK of MEDI-575 After the First Dose: Dose-normalized Maximum Serum Concentration (Cmax/Dose)
Description: The Cmax/dose after the first dose of MEDI-575 was obtained directly from the measured concentration-time curves. The concentration-time curve is the result of blood sampling at specified time points and its measured concentration of MEDI-575.
Time Frame: as for outcome 7
Population: All the participants who received first dose of MEDI-575 and for whom PK blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: μg/mL/mg
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 0.5 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 3 | 6 | 6
μg/mL/mg | 0.292 (0.0404) | 0.402 (0.125) | 0.335 (0.107) | 0.638 (0.171) | 0.655 (0.191) | 0.360 (0.0908) | 0.259 (0.0614) | 0.262 (0.0294) | 0.372 (0.103) | 0.357 (0.112)

10. Secondary Outcome: PK of MEDI-575 After the First Dose: Trough Serum Concentration (Ctrough)
Description: The Ctrough ie, measured concentration at the end of a dosing interval (taken directly before next dose administration) of MEDI-575 was obtained directly from the measured concentration-time curves. The concentration-time curve is the result of blood sampling at specified time points and its measured concentration of MEDI-575.
Time Frame: as for outcome 7
Population: All the participants who received first dose of MEDI-575 and from whom PK blood samples were collected and evaluated. Excluded participants were for whom it cannot be calculated (either number of doses received was less than 2 or standard deviation equals 0.000) or where dosing interval is more than 7 days or samples only collected up to 14 days.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 0.5 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 4
μg/mL | 8.97 (2.85) | 41.5 (13.8) | 72.6 (35.3) | 144 (18.0) | 199 (55.3) | 85.4 (40.8) | 223 (25.2) | NA (NA) — The mean was below limit of quantification and standard deviation cannot be calculated. | 59.0 (4.14) | 74.9 (22.6)

11. Secondary Outcome: PK of MEDI-575 After the First Dose: Area Under the Serum Concentration-time Curve Over the Dosing Interval (AUCτ)
Description: The AUCτ was obtained directly from the measured concentration-time curves. The concentration-time curve is the result of blood sampling at specified time points and its measured concentration of MEDI-575.
Time Frame: as for outcome 7
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: μg·day/mL
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 0.5 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 4
μg·day/mL | 201 (12.5) | 524 (166) | 835 (339) | 1870 (277) | 2080 (205) | 5100 (275) | 8340 (372) | 25.3 (7.69) | 763 (144) | 3760 (625)

12. Secondary Outcome: PK of MEDI-575 After the First Dose: Dose-normalized Area Under the Serum Concentration-time Curve (AUCτ/Dose)
Description: The AUCτ/dose was obtained directly from the measured concentration-time curves. The concentration-time curve is the result of blood sampling at specified time points and its measured concentration of MEDI-575.
Time Frame: as for outcome 7
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: μg·day/mL/mg
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 0.5 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 4
μg·day/mL/mg | 0.804 (0.0392) | 1.36 (0.441) | 1.19 (0.437) | 2.01 (0.418) | 2.12 (0.442) | 2.78 (0.767) | 2.35 (0.464) | 0.607 (0.197) | 1.15 (0.281) | 2.70 (0.438)

13. Secondary Outcome: Number of Participants Positive for Anti-drug Antibodies Formation for MEDI-575 at Any Visit
Description: Blood samples for immunogenicity assessments were collected from participants prior to the initiation of infusion of each treatment cycle of MEDI-575. Anti-MEDI-575 antibodies were analyzed using the electro-chemiluminescence (ECL) based method. Only the number of participants positive for anti-MEDI-575 antibodies at any visit are presented.
Time Frame: Preinfusion on Cycle 1 Day 1 and 30 days after the last dose, up to 112 weeks
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 6 | 6
Participants
  CYCLE 1 DAY 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  30 DAY POST | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response rate is defined as the proportion of participants with confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after the initial documentation of response. The CR is defined as disappearance of all target and non-target lesions, and normalization of tumor marker level. The PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: From study entry through the end of the study, up to 34 months
Population: Efficacy evaluable population: All participants who have received any treatment of MEDI-575 and at least one tumor assessment after the initiation of MEDI-575.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4
Percentage of participants | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 60.2]

15. Secondary Outcome: Time to Response
Description: Time to response was measured from the start of treatment with MEDI-575 to the first documentation of objective response (confirmed CR or PR). The time to response is assessed only for the participants who have achieved the objective response.
Population: Efficacy evaluable population with an objective response. Time to response was not estimable as there were no participants with an objective response.
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression. Disease progression is defined according to RECIST guidelines (ie, at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions). The duration of response was censored on the date of last tumor assessment documenting absence of disease progression for participants who have no documented progression prior to data cutoff, dropout, or the initiation of alternate anticancer treatment. Duration of response was calculated for the subgroup of participants with an objective response.
Population: Efficacy evaluable population with an objective response. Duration of response was not estimable as there were no participants with an objective response.
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) is defined as time from the start of treatment with MEDI-575 until the documentation of disease progression. Disease progression is defined according to RECIST guidelines (ie, at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions). The TTP was censored on the date of last tumor assessment documenting absence of tumor progression for participants who have no documented progression prior to data cutoff, dropout, or the initiation of alternate anticancer treatment. TTP was censored on the first date of treatment for the participants with no tumor assessments after the start of MEDI-575 treatment.
Time Frame: Start of treatment with MEDI-575 until the documentation of disease progression, up to 24 months
Population: Efficacy evaluable population. N= number of participants analyzed for this outcome measure
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 4
Months | 1.8 [1.5 to 24.8] | 1.4 [1.2 to NA] — The upper limit was not estimable | 1.2 [0.5 to NA] — The upper limit was not estimable | 1.4 [1.4 to 1.4] | 5.0 [1.2 to 8.8] | 2.9 [1.4 to 2.9] | 1.2 [1.0 to 1.4] | 1.4 [1.3 to 2.9] | 1.3 [1.2 to 5.7]

18. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as time from the start of treatment with MEDI-575 until the documentation of disease progression or death due to any cause, whichever occurred first. Disease progression is defined according to RECIST guidelines (ie, at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions). PFS was censored on the date of last tumor assessment documenting absence of tumor progression for participants who have no documented progression and were still alive prior to data cutoff, dropout, or the initiation of alternate anticancer treatment. PFS was censored on the first date of treatment for the participants with no tumor assessments after the start of MEDI-575 treatment.
Time Frame: Start of treatment with MEDI-575 until the documentation of disease progression or death due to any cause whichever occurs first, up to 24 months
Population: Efficacy evaluable population. N= number of participants analyzed for this outcome measure
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 4
Months | 1.8 [1.5 to 24.8] | 1.4 [1.2 to NA] — The upper limit was not estimable | 1.2 [0.5 to NA] — The upper limit was not estimable | 1.4 [1.4 to 1.4] | 5.0 [1.2 to 8.8] | 2.9 [1.4 to 2.9] | 1.2 [1.0 to 1.4] | 1.4 [1.3 to 2.9] | 1.3 [1.2 to 5.7]

19. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from the start of treatment with MEDI-575 until death. For the participants who were alive at the end of study or lost to follow-up, OS was censored on the last date when participants were known to be alive.
Time Frame: From the start of treatment with MEDI-575 until death or end of study, up to 33 months
Population: Efficacy evaluable population. N= number of participants analyzed for this outcome measure
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) | MEDI-575, 9.0 mg/kg QWk Expansion Phase | MEDI-575, 25 mg/kg Q3Wk Expansion Phase
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 3 | 2 | 2 | 4
Months | 9.0 [3.5 to NA] — The upper limit was not estimable | 3.7 [3.6 to 9.0] | 17.2 [7.4 to 27.0] | 5.5 [3.5 to 14.1] | 19.4 [3.4 to NA] — The upper limit was not estimable | 8.7 [1.8 to 10.5] | 10.3 [1.8 to NA] — The upper limit was not estimable | 5.4 [2.6 to NA] — The upper limit was not estimable | 5.9 [2.4 to 15.3]

ADVERSE EVENTS:
Time Frame: From the start of study drug administration through 30 days after last dose of MEDI-575, up to 112 weeks
Description: For treatment arms 9 mg/kg QWk and 25 mg/kg Q3Wk, both Escalation and Expansion Phase data are presented together for the Serious Adverse Events and Other Adverse Events.
Groups:
- MEDI-575, 9.0 mg/kg QWk Escalation/Expansion Phase (Cohort 3): MEDI-575 administered at 9.0 mg/kg as a 60-minute IV infusion on Study Days 1, 8, and 15 (QWk) of each 21 day treatment cycle until unacceptable toxicity, documentation of disease progression, or other reasons for participant withdrawal occurred.
- MEDI-575, 25 mg/kg Q3Wk Escalation/Expansion Phase (Cohort 6): MEDI-575 administered at 25.0 mg/kg as a 90-minute IV infusion on Study Day 1 of each 21-day treatment cycle (Q3Wk) until unacceptable toxicity, documentation of disease progression, or other reasons for participant withdrawal occurred.
Arm/Group | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) | MEDI-575, 9.0 mg/kg QWk Escalation/Expansion Phase (Cohort 3) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) | MEDI-575, 25 mg/kg Q3Wk Escalation/Expansion Phase (Cohort 6) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7)
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 8/11 | 0/3 | 0/3 | 2/9 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 10/11 | 3/3 | 3/3 | 9/9 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) (N=3) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) (N=3) | MEDI-575, 9.0 mg/kg QWk Escalation/Expansion Phase (Cohort 3) (N=11) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) (N=3) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) (N=3) | MEDI-575, 25 mg/kg Q3Wk Escalation/Expansion Phase (Cohort 6) (N=9) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) (N=3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-575, 3.0 mg/kg QWk Escalation Phase (Cohort 1) (N=3) | MEDI-575, 6.0 mg/kg QWk Escalation Phase (Cohort 2) (N=3) | MEDI-575, 9.0 mg/kg QWk Escalation/Expansion Phase (Cohort 3) (N=11) | MEDI-575, 12 mg/kg QWk Escalation Phase (Cohort 4) (N=3) | MEDI-575, 15 mg/kg QWk Escalation Phase (Cohort 5) (N=3) | MEDI-575, 25 mg/kg Q3Wk Escalation/Expansion Phase (Cohort 6) (N=9) | MEDI-575, 35 mg/kg Q3Wk Escalation Phase (Cohort 7) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 1 (4) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 2 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 4 (6) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (4) | 5 (6) | 2 (2) | 0 (0) | 6 (9) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (4) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 2 (10) | 2 (6) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (7) | 1 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.